CLINICAL TRIAL: NCT00250484
Title: The Effect of 10-Day Treatment of Repetitive Transcranial Magnetic Stimulation on Abdominal Pain in Patients With Chronic Pancreatitis
Brief Title: TMS Treatment for Pain in Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven Freedman, MD PhD Professor Medicine Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005P-000259 DK71851; R03DK071851 (NIH); NCT00130052 (obsolete NCT alias)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Idiopathic Chronic Pancreatitis; Pain
Keywords: analgesia; electric stimulation therapy; electric stimulation; pain; safety
MeSH Terms: conditions — Pain; Agnosia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (Active Comparator): Active treatment with TMS for 10 days.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Patients will receive no active TMS/treatment.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 1Hz transcranial Magnetic Stimulation for 10 days for 26 minutes each day
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Sham procedure of transcranial Magnetic Stimulation for 10 days for 26 minutes each day
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
The researchers aim to study the effects of repetitive transcranial magnetic stimulation (rTMS) on chronic visceral pain in patients with idiopathic chronic pancreatitis.

DETAILED DESCRIPTION:
The purpose of this protocol is to investigate a possible novel treatment for intractable visceral pain in patients with chronic pancreatitis. Pain is a major contributor to the poor quality of life in patients with chronic pancreatitis. The refractory nature of this condition to medical and surgical procedures prompted us to hypothesize that one mechanism leading to pain in these patients is the dysfunction of brain cortical regulation of visceral sensation. This notion is particularly supported by findings that patients with chronic pancreatitis can continue to experience disabling pain even after total pancreatectomy. This suggests that symptoms are sustained by a pancreas-independent, neural-based mechanism. Visceral sensation is particularly processed in the secondary somatosensory area - SII. Therefore, chronic pancreatitis pain may be sustained by a dysfunction of SII rather than by pancreatic inflammation alone. The researchers hypothesize further that the dysfunction of SII is one of hyper-excitability. According to this hypothesis, suppression of SII activity may help control the pain in patients with chronic pancreatitis. Temporary inhibition of SII activity can be obtained by a novel tool, namely transcranial magnetic stimulation (TMS), which can suppress brain excitability non-invasively beyond the duration of the TMS if appropriate stimulation parameters are employed. In the initial sham controlled, double blind pilot trial of 5 subjects with idiopathic chronic pancreatitis, TMS applied to SII resulted in significant pain improvement in 3 of the subjects. The researchers will rigorously test the hypothesis that chronic pancreatitis pain is sustained by a dysfunction of SII characterized by hyperexcitability through two specific aims:

1. The first aim of this study is to examine whether slow repetitive TMS (rTMS) applied to SII in patients with pain and chronic pancreatitis has an analgesic effect as measured by changes in the Visual Analogue Scale (VAS) for pain and a decrease in analgesic intake, as well as an overall improvement in quality of life. In addition, if this study finds a significant effect of rTMS on pain reduction, the duration of this effect will be further assessed. TMS will be applied at parameters of stimulation known to decrease excitability.
2. The second aim of the study is to assess the safety of rTMS in this patient population. In the pilot study none of the patients experienced any adverse effects of a single session of rTMS. However, the extension of the study protocol to a 10-day course of daily rTMS requires careful safety assessment. Fifteen-day courses of rTMS have been used for treatment of various neuropsychiatric diseases without any complications if safety guidelines are carefully followed. The researchers will adhere to the current safety recommendations for rTMS endorsed by the International Society for Transcranial Stimulation and the International Federation for Clinical Neurophysiology. Therefore, the researchers hypothesize that the proposed rTMS protocol will be safe for the patient population.
3. The third aim of the study is to study the physiologic mechanism of action of rTMS in these patients using magnetic resonance imaging (MRI). In doing so, the researchers aim to contribute to a better understanding of the pathophysiology of chronic pain in patients with pancreatitis by investigating the correlation between pain improvement and areas of brain activation. This could lead to the development of markers of therapeutic response. Magnetic resonance spectroscopy allows a non-invasive measure of GABAergic and glutamatergic activity in a defined volume of interest in the brain. The researchers hypothesize that the balance of GABA and glutamate will be abnormal in SII in patients with pain from chronic pancreatitis, with a relative decrease in GABA and increase in glutamate indicating an abnormal, hyperexcitable dysfunction. This abnormality will be normalized by rTMS in correlation with its analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible if:

They are age 18 years or older They have daily abdominal pain for at least three months attributed to their chronic pancreatitis Average pain scores (VAS) in the baseline period higher than 4.

The diagnosis of chronic pancreatitis will be based on the existence of chronic abdominal pain and at least one of the four following criteria:

Calcifications throughout the pancreas on plain abdominal radiograph. Endoscopically derived pancreatogram showing ductal changes consistent with chronic pancreatitis.

Abnormal secretin pancreatic function test with a peak bicarbonate level of less than 70 mEq/L (normal being >80 mEq/L).

Tissue diagnosis of chronic pancreatitis from a surgical specimen.

Exclusion Criteria:

Other causes of chronic pancreatitis will be excluded as follows:

Hereditary pancreatitis based on genetic mutations or a family history of pancreatitis; Alcohol abuse (the criteria for "at risk" [heavy] drinking established by the National Institute on Alcohol Abuse and Alcoholism [NIAAA], which suggest that the person is at risk for adverse consequences, are greater than 14 drinks per week or 4 drinks per occasion for men, and greater than 7 drinks per week or 3 drinks per occasion for women);

Medications associated with the development of pancreatitis (e.g. valproic acid, metronidazole, tetracycline, sulfonamides, nitrofurantoin, azathioprine, pentamidine), trauma, metabolic causes including hyperlipidemia and hypercalcemia, and autoimmune pancreatitis.

Participants will be excluded if there are known complications of chronic pancreatitis requiring interventions including pseudocysts or pancreatic duct obstruction or if there is the presence of cancer.

In addition, in order to minimize the risk of TMS, the following exclusion criteria will be followed:

Patients with a clinical diagnosis of severe depression including suicidal ideation; Prior neurosurgical procedure; Past history of epilepsy or family history of epilepsy; Previous head injury; Metal located in the head, i.e. shrapnel, surgical clips, or fragments from welding; Signs of increased intracranial pressure; Stroke; Chronic treatment with epileptogenic medications; Abnormal neurological examination other than as signs of the condition studied in the present protocol; Implanted pacemaker; Medication pump; Vagal stimulator; Deep brain stimulator; Transcutaneous electrical stimulation (TENS) unit and ventriculo-peritoneal shunt; Pregnancy; Other chronic medical conditions and history of substance abuse; History of medical and surgical therapies for pain within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Freedman, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan in protocol to share individual data

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 23 participants were recruited for the study, only 17 participated. This discrepancy is a result of 6 participants consenting for a realized exclusion criteria including a history of substance abuse or inability to commit.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.11 (11.27) | 46.71 (13.03) | 43.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Pain (Visual Analog Scale, CGI, PGA)
Description: Pain intensity and therefore changes in pain intensity were assessed using a 0-10 Visual Analog Scale where 0 represents the least amount of pain and 10 is the most pain imaginable. The pain evaluation was carried out by a blinded rater based off 1) baseline evaluation: 3 week long pain logs and a diary of pain medication intake, 2) treatment evaluations: participants were also asked to fill out daily pain logs following each TMS session and to keep a diary of pain medications during the CRC stay for the TMS course and 3)follow-up evaluation: finally, there was a follow up measurement 3 weeks after treatment.
Time Frame: 1 year
Measure: Number; unit: number of participants w/ reduced pain
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9 | 8
number of participants w/ reduced pain | 7 | 0

2. Secondary Outcome: Cognitive Assessment - Neuropsychological Battery
Description: Beck Depression Inventory (BDI), and Visual Analog Scale (VAS) for anxiety were assessed in subjects both as a baseline score before treatment was initiated as and upon conclusion of treatment.
  BDI is a 0-63 scale increasing with depression severity. A score from 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression, and 28-63 indicates severe depression. Higher values represent a worse outcome.
  VAS is a pain assessment ranging from 0-10 increasing with pain severity. High values represent a worse outcome.
Time Frame: Baseline and end of treatment at approximately 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 9 | 8
units on a scale
  BDI Beck Depression Inventory(baseline) | 23.05 (12.55) | 22.11 (10.71)
  BDI Beck Depression Inventory (after treatment) | 18.31 (10.54) | 21.69 (12.19)
  VAS Visual Analog Scale (baseline) | 4.26 (2.7) | 6.07 (1.66)
  VAS Visual Analog Scale(after treatment) | 3.35 (2.27) | 7.13 (2.90)

3. Secondary Outcome: Medication Use (Medication Diary)
Description: Data was not collected or recorded because this outcome measure was no longer considered useful or relevant in the study.
Time Frame: Baseline and end of treatment at approximately 1 year
Population: Data was not collected. Data was not collected or recorded because this outcome measure was no longer considered useful or relevant in the study.
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse data were collected up to 30 minutes after rTMS. Adverse effects were assessed using a structured questionnaire listing the most common adverse effects associated with TMS.
Description: Headache, neck pain, scalp burning, hearing difficulties, cognitive changes, changes in concentration, and/or mood changes were assessed.
Arm/Group | Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/9 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Magnetic Stimulation (N=9) | Sham Transcranial Magnetic Stimulation (N=8)
Headache (Nervous system disorders) | 4 (41) | 2 (19)
Neck (Nervous system disorders) | 2 (18) | 1 (3)
Scalp (Nervous system disorders) | 1 (5) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0)
Hearing (Nervous system disorders) | 1 (2) | 0 (0)
Cognition (Nervous system disorders) | 2 (15) | 1 (13)
concentration (Nervous system disorders) | 2 (29) | 2 (30)
mood (Nervous system disorders) | 2 (21) | 2 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No